CLINICAL TRIAL: NCT04928547
Title: An Integrated System for the Assessment of Carotid Plaque Stability Based on the Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-460-1
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Carotid Plaque Stability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- U.S.
  Interventions: Diagnostic Test: Test
- MRI
  Interventions: Diagnostic Test: Test

INTERVENTIONS:
Diagnostic Test: Test — Different test

SUMMARY:
The project will be properly embedded in the clinical practice landscape to both provide a real-world context for research requirements gathering and research result assessment, and a practical application context from the industrial perspective. The landing is planned for cardiology solutions as carotid plaque assessment that can be value-adding features to tackle the current challenges of stroke prediction. The development of stroke prediction model could accelerate the R&D process and land to key market ultrasound prototypes/products in an agile way. Collaboration and alignment with key market business and R&D (China Digital Innovation CDI) through workshops and hackathons will be a unique feature of this agile project.

DETAILED DESCRIPTION:
Stroke is a global disease with high mortality and disability. Evaluation of the stability of carotid plaque has important clinical significance for stroke prevention.

As a practical, fast, non-invasive, non-radiative inspection technique, ultrasound is widely used in the evaluation of carotid plaque stability. There are many methods for evaluating the stability of carotid plaque by ultrasound. The texture features extracted from two-dimensional ultrasound images can be used to quantify subtle differences in follow up scanning. The elastography of the plaques can be used to quantify changes in the elastic properties of reactive plaques. Contrast enhanced ultrasound (CEUS) can be used to quantify the density of microvessels. However, the results obtained by these different methods are biased and show poor agreement. We lack a unified, systematic evaluation system and objective guideline for plaque stability assessment. In this context, the topic of plaque stability assessment has been intensively explored by researchers from all over the world. Based on state-of-the-art assessment, we found that some plaques that were judged stable on ultrasound did eventually rupture. On the contrary, some unstable plaques on ultrasound did not cause stroke. This confusion indicates that plaque rupture is not only related to its intrinsic characteristics, such as size, shape, composition etc., but also to external factors such as biomechanics, strain, flow field, etc.. In order to achieve a better understanding of the pathological plaque behaviour, it is necessary to study the hemodynamic problems in the arteries, such as wall shear stress, flow separation, and secondary flow. The recent rapid developments in artificial-intelligence techniques have been widely used in medical imaging and image analysis. These techniques allow supervised learning taking full advantage of the available big data. Therefore, the main purpose of this study is to use artificial intelligence technique to i) evaluate a number of indicators including plaque histology, hemodynamics, etc., ii) establish a uniform and quantitative criteria for judging the stability of carotid plaque.

The key scientific problem to be solved in this project is to establish an objective model for predicting the risk of carotid plaque rupture for clinical decisionmaking.

It can be mainly divided into three main modules: database establishment, model training and clinical validation.

1. Database establishment

1. Obtaining clinical information of the patients from the electronic medical record system.
2. Use of image analysis techniques in ultrasound images to study the relationship between different image texture parameters and plaque histological composition. A method for evaluating the stability of carotid plaque based on texture parameters will be established.
3. Use of ultrasound (shear-wave) elastography to establish a method for assessing the carotid-plaque vulnerability based on the assessment of tissue elasticity.
4. Combining carotid velocity vector imaging with the blood-flow vortex manipulation technique to achieve an accurate measurement of the central position of the vulnerable plaque blood flow vortex and the orbital angular momentum, providing a new technique for vulnerable plaque detection based on vortex vector blood flow. Block detection new technology. The biomechanical characteristics of arterial plaques will be evaluated by detecting the synchrony and coordination of the arterial wall. The relationship between the biomechanical characteristics and stability of different types of plaques in the cardiac cycle will also be investigated.
5. Use of quantitative CEUS analysis and localization microscopy to study the relationship between CEUS and neovascularization in carotid plaques, focusing on the influence of microvessel density, architecture, and other quantitative features extracted from CEUS. Based on these features, a prediction model for plaque rupture will be designed and evaluated.
6. Use of computational fluid dynamics modeling to study the effects of geometrical changes on local hemodynamics and blood component concentration distribution during plaque growth. Further analysis of the growth mechanism of plaque and its effect on hemodynamics will be made.

2. Deep-learning model After obtaining all the parameters mentioned above, the correlation between these parameters and carotid plaque stability will be studied through machine learning.

A machine-learning classifier will be designed that takes the extracted features as input. Feature selection will be implemented through k-fold cross-validation to identify the set of complementary features that most contribute to assess plaque stability and predict plaque rupture. In particular, we aim at predicting whether a stroke will occur within 1 year. When sufficient data is available, a deep convolutional neural network will also be designed and trained to learn the prediction model. In this process, the risk of overfitting will be carefully considered by evaluating the classification performance over training, test, and validation sets.

As a result, the model complexity will be adjusted to the available training sets.

3. clinical evaluation The validation of the developed stroke prediction model from rupture of carotid plaques will be extended to a number of hospitals. The model reliability and usability will be tested. Model update and improvement is envisaged in a cyclic fashion, profiting from clinical results and feedback. The accuracy rate auxiliary decision support is expected to levels that are not lower than 90%.

ELIGIBILITY:
Inclusion Criteria:

1. Age is greater than or equal to 18 years old and less than or equal to 80 years old;
2. At least one imaging examination suggests the presence of carotid artery plaque;
3. No allergy and other contraindications to ultrasound contrast;
4. Contrast-enhanced ultrasound examination of carotid artery plaque is required;
5. Volunteer to join this research project and sign informed consent.

Exclusion Criteria:

1. Patients who are unable to coordinate their body position or hold their breath during the ultrasound examination;
2. Patients with severe lack of clinical data;
3. During the follow-up, use drugs for the treatment of carotid plaque except lipid-lowering drugs, antiplatelet drugs, antioxidants, and calcium channel blockers;
4. Follow up those who have lost contact;
5. Ischemic stroke caused by non-carotid artery plaque shedding;
6. Patients with atrial fibrillation and other serious heart diseases;
7. A history of allergy to ultrasound contrast agents.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: According to previous research and experience, the percentage of neovascularization grade II and above accounted for about 79% of all plaques in the enrolled patients, neovascularization grade I accounted for 21%, neovascularization grade II predicted the recurrence of stroke in the same basin 10%, neovascularization I The recurrence rate of stroke in the same watershed below grade is 6%, and the sample size is calculated to be about 100 cases. Gray-scale ultrasound shows the presence or absence of hypoechoic and iso-echoic, calcified nodules and other characteristics. The loss to follow-up rate is calculated as 10-15%. This study intends to include 2000 patients with acute anterior circulation ischemic stroke. A total of 100 patients were enrolled in this research center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Stroke | 3 years